CLINICAL TRIAL: NCT06131944
Title: Prevention Strategies to Enhance Young Children's Sleep Development - Part 1
Brief Title: A Combined School- and Home-Based Sleep Promotion Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Sarah Burkart, Assistant Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00125230; 5P20GM130420 (NIH)
Record Dates: First submitted 2023-10-11; First posted 2023-11-15 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rested & Ready to Learn (Experimental): All participants will receive the four-week Rested & Ready to Learn sleep promotion program which includes text messaging to parents, home activities for parents and children to complete together, and brief classroom lessons.
  Interventions: Behavioral: Rested & Ready to Learn

INTERVENTIONS:
Behavioral: Rested & Ready to Learn — The intervention arm targets improving young children's sleep by providing parents with sleep education and activities to do at home with their child. Classroom teachers will also deliver a brief lesson aligned with intervention topics to reinforce key messaging in the classroom. The sleep intervention will focus on the benefits of sleep (physical health, social-emotional health, classroom participation/learning), creating and sticking to a bedtime routine, screen use before bed, and developmentally appropriate sleep behavior.

SUMMARY:
The goal of this single group trial is to test the feasibility and acceptability of a combined school- and home-based sleep promotion program for young children prior to the kindergarten transition.

DETAILED DESCRIPTION:
This single group pilot study will test a combined school- and home-based sleep promotion intervention designed to improve young children's sleep and classroom behavior. All participants will receive the intervention. Intervention content will be delivered via text message to parents' phones and in the classroom. The primary aim of this study is to assess the feasibility and acceptability of the intervention. The secondary aim is to assess the preliminary signal of effect on children's sleep and classroom behavior. Findings from this study will inform any necessary intervention modifications prior to a pilot randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Child between the ages of 4-6 years
* Currently enrolled in a participating school's 4-year-old kindergarten (4K) classroom
* Parent/guardian willing to complete questionnaires in English
* Parent/guardian must have access to a mobile phone with texting capability

Exclusion Criteria:

* Parent or child has a medical condition that impairs their ability to participate

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Trial-related feasibility - recruitment capability | Through recruitment period, up to 6 weeks
  Recruitment capability will be measured by the proportion of eligible children who enroll at baseline.
Trial-related feasibility - retention | Weekly through study completion (weeks 1-5)
  Retention will be measured by the proportion of enrolled children who remain in the study through the length of the intervention. Reasons for dropout will also be assessed.
Intervention-related feasibility - intervention fidelity | Weekly through study completion (weeks 1-4)
  Intervention fidelity, the delivery of the intervention as originally planned, will be assessed via teacher report. Intervention fidelity will be assessed with a study-specific questionnaire to assess if all classroom components were delivered as planned.
Intervention-related feasibility - rate of attendance | Weekly through study completion (weeks 1-4)
  Children's attendance at school during intervention sessions will be provided by class records.
Intervention-related feasibility - participant adherence to intervention (home) | Weekly through study completion (weeks 1-4)
  Adherence to the home-based component will rely on link usage data to assess parent engagement with the online materials. Investigators will extract information related to the number of parents who click links from weekly material and number of parents who do not open links.
Intervention-related feasibility - participant adherence to intervention (school) | Weekly through study completion (weeks 1-4)
  School-based adherence will be assessed by a teacher-completed survey which will indicate whether or not they implemented the intervention each week.
Intervention-related feasibility - data collection completion rates | Weekly through study completion (weeks 1-4)
  Data collection completion rates will be calculated to understand the feasibility of data collection protocols.
Intervention-related feasibility - data collection feasibility | Post-intervention (week 5-7)
  Feasibility of data collection procedures will be assessed with qualitative feedback from parents during semi-structured interviews following the study.
Acceptability | Weekly through study completion (weeks 1-4), post-intervention (week 5-7)
  Acceptability of the intervention conditions is defined as participants' perception that the intervention is satisfactory and will be assessed with short weekly questionnaires for parents and teachers. Overall acceptability will be assessed with an exit-survey consisting of Likert-scale items and open-ended responses to understand likes/dislikes, content, logistics, and feedback for future iterations. Likert-style questions will have response options ranging from 1-5 with greater scores representing higher acceptability.

SECONDARY OUTCOMES:
Child sleep - device-based duration | Baseline (week 0) and post-intervention (week 5)
  Objective nocturnal sleep duration will be assessed using Axivity AX3 accelerometers worn on the non-dominant wrist for 7 days. Raw accelerometry data will be processed with open-source software, GGIR.
Child sleep - device-based timing | Baseline (week 0) and post-intervention (week 5)
  Objective sleep timing will be assessed using Axivity AX3 accelerometers worn on the non-dominant wrist for 7 days. Raw accelerometry data will be processed with open-source software, GGIR.
Child sleep - Bedtime Routines Questionnaire | Baseline (week 0) and post-intervention (week 5)
  Parents will complete the Bedtime Routines Questionnaire which contains 31 items on a 5-point Likert scale. This questionnaire results in two subscales - bedtime routine consistency and routine behaviors and environment. Higher scores indicate more consistent bedtime routines.
Child behavior | Baseline (week 0) and post-intervention (week 5)
  Parents and teachers will complete the Child Self-Regulation and Behavior Questionnaire (CSBQ, ~10 min) which contains 34 items describing children's typical self-regulation and social behaviors in the home (parent version) and classroom (teacher version). Respondents describe what the child's behavior is like on a five-point scale ranging from "Not true" to "Very true." The CSBQ provides the following subscales: self-regulation, sociability, externalizing problems, internalizing problems, and prosocial behavior. The CSBQ is valid and reliable in children ages 3-6 years.
Child inhibition | Baseline (week 0) and post-intervention (week 5)
  Inhibition (i.e., the ability to control behavioral impulses) will be assessed with the Go/No-Go task in which children are asked to identify fish and avoid sharks shown on the screen on an iPad as part of the freely accessible Early Years Toolbox. An impulse control score is calculated (% Go Accuracy x % No-Go Accuracy), which reflects the child's ability to withhold their response in the context of the strength of that typical (pre-potent) response.
Child working memory | Baseline (week 0) and post-intervention (week 5)
  Working memory (i.e., amount of information that can be coordinated in the mind) will be assessed with the Mr. Ant task in which children will recall and identify the location of colorful stickers on Mr. Ant's body on an iPad as part of the freely accessible Early Years Toolbox. For the Mr Ant task, scores are calculated using a point score calculated as: beginning from level 1, one point for each consecutive level in which at least two of the three trials were performed accurately, plus 1/3 of a point for all correct trials thereafter.
Child cognitive flexibility | Baseline (week 0) and post-intervention (week 5)
  Cognitive flexibility (i.e., the ability to control and redirect attention) will be assessed with the Card Sorting task in which children will sort cards by color and then shape on an iPad as part of the freely accessible Early Years Toolbox. For the Card Sorting task, investigators tend to review the accuracy of Block 1 (pre-switch) and Block 2 (post-switch). Since a post-switch accuracy score intends to index the extent to which a child could successfully switch from one sorting rule to the next, investigators will swap the two scores if the post-switch accuracy is larger than the pre-switch accuracy. This ensures that final post-switch scores (Block 2 + Block 3) reflects the child's ability to successfully switch between sorting rules.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Burkart, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No